CLINICAL TRIAL: NCT06684834
Title: The Effects of Intermittent Carbohydrate Restriction on Metabolic Health and Energy Balance in Adults with Abdominal Overweight and Obesity
Brief Title: Intermittent Carbohydrate Restriction in Cardiometabolic Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Bath (Other)
Responsible Party: Principal Investigator, Guoda Karoblyte, Principal Investigator, University of Bath
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 323721
Record Dates: First submitted 2024-10-24; First posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Obesity and Overweight
Keywords: carbohydrate restriction; carbohydrate timing; intermittent carbohydrate restriction; intermittent energy restriction; evening carbohydrate restriction; carbohydrate periodisation
MeSH Terms: conditions — Obesity; Overweight

STUDY DESIGN:
Intervention Model Description: A randomised, three-arm parallel-group study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 5:2 carbohydrate restriction (5:2CR) (Experimental): Laboratory measurements will be obtained before and after the intervention. Physical activity, dietary intake and interstitial glucose concentrations will be monitored in free-living conditions throughout the intervention.
  Interventions: Other: 5:2 carbohydrate restriction
- Early time-restricted carbohydrate intake (eTRC) (Experimental): Laboratory measurements will be obtained before and after the intervention. Physical activity, dietary intake and interstitial glucose concentrations will be monitored in free-living conditions throughout the intervention.
  Interventions: Other: Early time-restricted carbohydrate intake
- Lifestyle maintenance (control) (No Intervention): Laboratory measurements will be obtained before and after the intervention. Physical activity, dietary intake and interstitial glucose concentrations will be monitored in free-living conditions throughout the intervention.

INTERVENTIONS:
Other: 5:2 carbohydrate restriction — Carbohydrate ingestion restricted to <8% of energy intake on 2 self-selected consecutive days each week over 28-30 days. Ad libitum dietary amount, type and pattern followed on the remaining 5 days each week.
  Arms: 5:2 carbohydrate restriction (5:2CR)
Other: Early time-restricted carbohydrate intake — Carbohydrate intake restricted to <8% of energy intake after 4pm each day for 28 days. Ad libitum dietary amount, type and pattern followed before 4pm.
  Arms: Early time-restricted carbohydrate intake (eTRC)

SUMMARY:
Metabolic conditions, such as heart disease, type 2 diabetes, and metabolic syndrome, are among the leading causes of disability and mortality worldwide. Identifying innovative lifestyle strategies to reduce metabolic risk remains a public health priority. Further research is essential to understand how low carbohydrate intake influences human metabolism and how intermittent carbohydrate restriction impacts weight loss and metabolic health markers.

This study will investigate two interventions that restrict dietary carbohydrate intake on different schedules, examining their effects on metabolic health and energy balance in adults with abdominal overweight or obesity. The physiological mechanisms potentially underlying these effects will be explored by measuring a range of lifestyle and metabolic health parameters in both free-living and laboratory settings. A digital behaviour-change intervention will be incorporated after the dietary intervention to assess whether any metabolic effects can be sustained over time.

The study employs a three-arm parallel-group design consisting of a two-week lifestyle monitoring phase, a four-week dietary intervention, and a four-week digital intervention, with four laboratory visits throughout each phase. During the dietary intervention, participants will be allocated to one of three groups: (i) carbohydrate restriction (<8% of energy intake) on two consecutive days per week, (ii) carbohydrate restriction after 4 pm each day, or (iii) no dietary changes.

Dietary intake, physical activity, and glucose levels will be monitored through wearable devices in free-living conditions. The digital intervention will use a mobile health application that provides individualised lifestyle recommendations and education based on data collected in free-living conditions. Laboratory-based measures will include anthropometry, body composition scans, indirect calorimetry, blood pressure monitoring, fat biopsies, and postprandial sampling of blood and expired air.

ELIGIBILITY:
Inclusion Criteria:

1. Waist circumference of ≥94 cm (37 inches) if male and ≥80 cm (31.5 inches) if female, or BMI above 25 kg/m2
2. Fat mass index (FMI) of >6 kg/m2 for males, and >9 kg/m2 for females
3. Aged between 18-65 years
4. Has maintained a stable weight in the last three months (<3% change in body mass)
5. Keeps track of menstrual cycle regularity or oral contraceptive use (females only)

Exclusion Criteria:

1. Has a body weight of ≥120kg
2. Plans to undertake other lifestyle modifications during the study to manage weight (e.g. changes in dietary intake or activity levels)
3. Current or previous eating disorder
4. Diagnosed with major chronic conditions (e.g. type 2 diabetes, coronary heart disease, cancer, chronic kidney disease, etc.)
5. Use of medication that may interfere with study outcomes (e.g. glucose or lipid lowering medications)
6. Currently or recently pregnant (within last 6 months), planning to get pregnant or currently lactating
7. Has donated more than 500ml of blood in the last 3 months prior to the initial laboratory visit
8. Insufficient mental capacity or language skills to independently understand and follow the study protocol
9. Dietary restrictions to ingredients in test meals (e.g. gluten and lactose)
10. Has an irregular sleeping pattern (e.g. due to undertaking night-shift work)
11. Any condition, concurrent intervention or behaviour deemed either to pose undue personal risk to the participant or to introduce bias into the experiment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-09-05 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2036-10 (Estimated)

PRIMARY OUTCOMES:
Post Prandial Triglyceride Area Under the Curve (AUC) | Pre and post intervention (4 weeks)
  Plasma triglyceride concentrations assessed postprandially for 5 hours after a mixed meal test

SECONDARY OUTCOMES:
Fat Mass | Pre and post intervention (4 weeks)
  Measured in kilogrammes using Dual Energy X-ray Absorptiometry
Lean Body Mass | Pre and post intervention (4 weeks)
  Measured in kilogrammes using Dual Energy X-ray Absorptiometry
Fasting and Post Prandial Glucose Concentration | Pre and post intervention (4 weeks)
  Plasma glucose concentrations assessed after an overnight fast, postprandially for 5 hours after a mixed meal test
Fasting and Post Prandial Insulin Concentration | Pre and post intervention (4 weeks)
  Plasma insulin concentrations assessed after an overnight fast, postprandially for 5 hours after a mixed meal test
Fasting and Post Prandial NEFA Concentration | Pre and post intervention (4 weeks)
  Plasma NEFA concentrations assessed after an overnight fast, postprandially for 5 hours after a mixed meal test
Fasting Triglyceride Concentration | Pre and post intervention (4 weeks)
  Plasma triglyceride concentrations assessed after an overnight fast
Fasting Total Cholesterol Concentration | Pre and post intervention (4 weeks)
  Assessed after an overnight fast
Fasting LDL-C Concentration | Pre and post intervention (4 weeks)
  Assessed after an overnight fast
Fasting HDL-C Concentration | Pre and post intervention (4 weeks)
  Assessed after an overnight fast
Substrate Oxidation | Pre and post intervention (4 weeks)
  Carbohydrate and fat oxidation rates will be measured using indirect calorimetry at rest and every hour postprandially
Adipose Tissue Gene Expression | Pre and post intervention (4 weeks)
  Expression of several genes related to energy metabolism in adipose biopsies using real-time polymerase chain reaction (RT-PCR)
Adipose Tissue Protein Expression | Pre and post intervention (4 weeks)
  Expression of several proteins related to energy metabolism in adipose biopsies using Western blot

OTHER OUTCOMES:
Physical Activity Energy Expenditure (kJ or kcal) | 1 week during baseline monitoring, and weeks 1 and 4 of the intervention
  Assessed using combined heart rate and accelerometery wearable monitor (Actiheart™) in free-living conditions.
Time Spent in Different Physical Activity Intensities (minutes) | 1 week during baseline monitoring, and weeks 1 and 4 of the intervention
  Assessed using combined heart rate and accelerometery wearable monitor (Actiheart™) in free-living conditions
Dietary Intake | 1 week during baseline monitoring, and weeks 1 and 4 of intervention
  Dietary records manually kept by study participants
Interstitial Glucose | 2 weeks during baseline monitoring, 2 weeks during weeks 3-4 of intervention
  Continuous glucose records will be used to capture interstitial glucose before and during the intervention
Sleep Quality | Pre and post intervention (10 weeks)
  Self-reported sleep quality will be assessed via the Pittsburgh Sleep Quality Index (PSQI) questionnaire, consisting of 9 questions. Seven component scores are derived, scored from 0 (no difficulty) to 3 (severe difficulty)
Diet Satisfaction | Pre and post intervention (10 weeks)
  Diet satisfaction will be assessed via the 28-item Diet Satisfaction Questionnaire (28-DSQ), scored on a five-point Likert scale with 1 being 'Disagree Strongly' and 5 being 'Agree Strongly'
Engagement with Mobile Application | 4 weeks post intervention
  Data on number of sessions, session length, session interval and session frequency will be obtained through the Salus Metabolism mobile health application
Usability of Mobile Application | 4 weeks post intervention
  Assessed via the mHealth App Usability Questionnaire, consisting of 16 statements scored on a seven-point Likert scale with 1 being 'Disagree' and 7 being 'Agree'
Subjective App Usability and Engagement | 4 weeks post intervention
  Participants will be asked to provide feedback on the Salus Metabolism mHealth application through a semi-structured interview. Thematic analysis will be used to analyse interview data.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bath, Bath, Somerset, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided